CLINICAL TRIAL: NCT01929226
Title: A Double-Blind, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of a Single Intravenous Dose of ETI-204 in Adult Volunteers
Brief Title: Safety, Tolerability, and PK of a Single Intravenous Dose of ETI-204 in Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elusys Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AH104
Record Dates: First submitted 2013-08-02; First posted 2013-08-27 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-01

CONDITIONS: Inhalational Anthrax
Keywords: anthrax, monoclonal antibody, ETI-204, safety, PK
MeSH Terms: conditions — Inhalation anthrax; Anthrax | interventions — obiltoxaximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ETI-204 (Experimental): A single intravenous dose of 16 mg/kg ETI-204 infused over 90 minutes on Day 1
  Interventions: Biological: ETI-204
- Placebo for ETI-204 (Placebo Comparator): A single intravenous dose of ETI-204-placebo infused over 90 minutes on Day 1
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ETI-204 — Monoclonal Antibody
  Arms: ETI-204
Other: Placebo — Placebo for ETI-204
  Arms: Placebo for ETI-204

SUMMARY:
To evaluate the safety and tolerability and pharmacokinetics (PK) of a single intravenous (IV) dose of ETI-204 in adult volunteers.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled study of a single IV dose of 16 mg/kg ETI-204 in adult volunteers (210 subjects ETI-204; 70 subjects placebo).

The total duration of the study for each subject will be approximately 100 days divided as follows:

Screening: Days -28 to -2; In-unit Phase: Day -1, Day 1, and Day 2; Out-of-unit Visits: Day 8 (±2 days); Day 15 (±3 days); Day 29 (±3 days); Day 43 (±3 days); Final Visit: Day 71 (±4 days).

Following completion of a screening visit subjects who qualify for entry into the study will be randomized to receive either ETI-204 or matching placebo on Day 1 in a 3:1 ratio. Subjects will be discharged from the clinic on Day 2 following completion of study assessments and will return for five additional visits on Days 8, 15, 29, 43 and 71.

The first 12 subjects will be dosed in groups of no more than 4 subjects/day. A blinded safety review of the available clinical and laboratory AE data up to and including Day 2 will be completed for the first 12 subjects before any additional subjects are dosed. This review will be conducted by the Investigator in conjunction with the Clinical Trial Steering Committee. If the outcome of this review is satisfactory, dosing of additional subjects will be permitted to continue and subjects may be dosed in group sizes larger than 4.

After Amendment 1, premedication with 50 mg oral diphenhydramine approximately 30 minutes prior to the start of study drug infusion was required.

ELIGIBILITY:
Inclusion Criteria:

1. Females or males ≥ 18 years of age
2. All females, regardless of childbearing potential, must have a negative serum beta human chorionic gonadotropin (β-hCG) pregnancy test at Screening and Day -1
3. Females of childbearing potential (i.e., not postmenopausal or surgically sterile) must agree to practice abstinence or to use a medically accepted method of contraception from the time of Screening through 30 days after final study visit. Acceptable methods of contraception include diaphragm with spermicide; sponge with spermicide; condom with spermicide; or intrauterine device with condom or spermicide. The following contraceptive methods are acceptable only when used with a condom and spermicide: birth control pills, birth control patches, vaginal ring, hormone under the skin, or hormone injections
4. Postmenopausal females, defined as females who have had amenorrhea for at least 12 months either naturally or following cessation of all exogenous hormonal treatments and have a follicle stimulating hormone (FSH) level of > 40 mIU/mL at Screening
5. Females who have undergone surgical sterilization, including hysterectomy, bilateral oophorectomy, bilateral salpingectomy, tubal ligation, or tubal essure
6. Males must agree to practice abstinence or use a condom with spermicide and refrain from sperm donation during the study and for 30 days after the final study visit
7. Provide written informed consent
8. Willing to comply with study restrictions

Exclusion Criteria:

1. Pregnant or lactating woman
2. Clinically significant comorbidity that would interfere with completion of the study procedures or objectives, or compromise the subject's safety
3. Seated systolic blood pressure (BP) ≥ 150 mmHg or ≤ 90 mmHg or diastolic BP ≥ 95 mmHg
4. Use of H1 receptor antagonists (i.e. antihistamines) within 5 days prior to Day 1
5. Evidence of drug or alcohol abuse as determined by the Investigator within 6 months of Day 1
6. Positive test result for drugs of abuse (with the exception of medically prescribed drugs) at Screening or on Day -1
7. Positive test for alcohol at Screening; exclusion is subject to the Investigator's discretion; subjects who test positive for alcohol at Day -1 are excluded from the study
8. Treatment with an investigational agent within 30 days of Day 1 or within five half-lives of the investigational agent at Day 1 (whichever is longer)
9. Congenital or acquired immunodeficiency syndrome
10. Prior solid organ or bone marrow transplant
11. Positive test for Hepatitis B (surface antigen), Hepatitis C, or human immunodeficiency virus (HIV) at Screening
12. History of prior treatment for anthrax exposure or prior anthrax infection
13. Prior immunization with any approved or investigational anthrax vaccine or prior treatment with an investigational anthrax treatment (i.e., ETI-204, raxibacumab, or anthrax immune globulin)
14. Military personnel deployed in 1990 or after, unless the subject can provide documentation demonstrating they have not previously received any approved or investigational anthrax vaccine
15. Use of systemic steroids, immunosuppressive agents, anticoagulants, or anti-arrhythmics within 1 year prior to Day 1. A single short course (i.e., less than 14 days) of systemic steroid therapy is allowed provided it concluded more than 6 months prior to Day 1
16. Donation or loss of > 500 mL of blood within 30 days or plasma within 7 days of Day 1
17. Prior stroke, epilepsy, relapsing or degenerative central nervous system disease, or relapsing or degenerative ocular disease
18. Myocardial infarction or acute coronary syndrome in the past 5 years, active angina pectoris, or heart failure (New York Heart Association scale > 1)
19. History of chronic liver disease
20. Calculated creatinine clearance (CrCl) of < 30 mL/min using the Cockcroft-Gault equation
21. Any clinically significant abnormality, in the Investigator's opinion, on electrocardiogram (ECG) or clinical laboratory tests (hematology, clinical chemistry, or urinalysis) at Screening; Out of range results may be repeated to confirm.
22. History of allergic or hypersensitivity reactions to other therapeutic antibodies or immunoglobulins
23. History of any malignant neoplasm within the last 5 years, with the exception of adequately treated localized or in situ non-melanoma carcinoma of the skin (i.e., basal cell carcinoma) or the cervix
24. Subjects who, in the opinion of the Investigator, are not suitable candidates for enrollment or who may not comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2013-07-09; Primary Completion 2013-11-29 (Actual); Study Completion 2013-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex King, MD, Principal Investigator — Covance; Lori Sieboldt, MD, Principal Investigator — Covance Clinical Research - Evansville, IN; Debra Mandarino, MD, Principal Investigator — Covance Research, Madison, WI; H. Frank Farmer, PhD, MD, Principal Investigator — Covance Research - Daytona Beach, Fl
Locations (1):
- Covance Clinical Research Inc., Dallas, Texas, United States

REFERENCES:
- [Derived] Nagy CF, Leach TS, Hoffman JH, Czech A, Carpenter SE, Guttendorf R. Pharmacokinetics and Tolerability of Obiltoxaximab: A Report of 5 Healthy Volunteer Studies. Clin Ther. 2016 Sep;38(9):2083-2097.e7. doi: 10.1016/j.clinthera.2016.07.170. Epub 2016 Aug 24. PMID 27568215

RESULTS

PARTICIPANT FLOW:
Groups:
- ETI-204: Intravenously (IV), single dose
  ETI-204: Monoclonal Antibody
- Placebo: Intravenously (IV), single dose
  Placebo: Placebo comparator
Period: Overall Study
Arm/Group | ETI-204 | Placebo
Started | 210 | 70
Completed | 205 | 69
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ETI-204 | Placebo | Total
Number analyzed (Participants) | 210 | 70 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (15.59) | 41.5 (13.90) | 42.2 (15.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 32 | 136
  Male | 106 | 38 | 144
Region of Enrollment [Number; unit: participants]
  United States | 210 | 70 | 280

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Adverse Events
Description: Safety was assessed for all subjects in the safety population by collecting and monitoring vital signs, clinical laboratory tests, ECGs, physical examinations, skin assessments, infusion site assessments, and adverse events.
Time Frame: Up to 71 days or 101 days (30 days after the final study visit) for subjects with ongoing adverse events at the final study visit, for each group.
Population: All randomized participants who received study drug.
Measure: Count of Participants; unit: Participants
Groups:
- ETI-204: Participants were administered a single intravenous (IV) infusion of 16 mg/kg ETI-204 in 0.9% sterile sodium chloride in a total volume of 250 mL over 90 minutes. ,
  Following a protocol amendment, 147(70%) participants were premedicated with 50 mg oral diphenhydramine approximately 30 minutes prior to the start of the infusion.
- Placebo: Participants were administered a single intravenous (IV) infusion of ETI-204 Placebo in 0.9% sterile sodium chloride in a total volume of 250 mL over 90 minutes. ,
  Following a protocol amendment, 48(68.6%) participants were premedicated with 50 mg oral diphenhydramine approximately 30 minutes prior to the start of the infusion.
Arm/Group | ETI-204 | Placebo
Number analyzed (Participants) | 210 | 70
Participants | 88 | 27

2. Secondary Outcome: Maximum Observed Plasma Concentration of ETI-204 (Cmax)
Description: Blood samples were obtained and serum concentrations were determined using a validated enzyme-linked immunosorbent assay method with an assay range of 100 ng/mL to 5000 ng/mL.
Time Frame: On Day 1, prior to the start of infusion, at the end of infusion, and 3 and 8 hours after the start of infusion and on Days 2, 8, 15, 29, 43, and 71.
Population: Of the 210 participants who received ETI-204, 202 were included in the PK population. One was excluded due to missing dosing record and 7 received partial doses of ETI-204 (6 discontinued study drug due to an AE and one received a partial dose because of mechanical issues with the infusion pump).
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- ETI-204: Participants were administered a single intravenous (IV) infusion of 16 mg/kg ETI-204 in 0.9% sterile sodium chloride in a total volume of 250 mL over 90 minutes. ,
  Following a protocol amendment, 147(70%) participants were premedicated with 50 mg oral diphenhydramine approximately 30
Arm/Group | ETI-204 | Placebo
Number analyzed (Participants) | 202 | 0
µg/mL | 400 (91.2) |

3. Secondary Outcome: Time to Maximum Observed Plasma Concentration of ETI-204 (Tmax)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | ETI-204 | Placebo
Number analyzed (Participants) | 202 | 0
days | 0.0782 [0.0674 to 1.01] |

4. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Time of Last Measurable Concentration (AUC0-last)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: Of the 210 participants who received ETI-204, 202 were included in the PK population. Reasons for exclusion were: missing dosing record (1), discontinued study drug due to an AE (6) and mechanical issues with the infusion pump (1). 3 additional participants were excluded from the AUC0-last calculation because of missing PK collection time points.
Measure: Mean (Standard Deviation); unit: µg.day/mL
Arm/Group | ETI-204 | Placebo
Number analyzed (Participants) | 199 | 0
µg.day/mL | 4770 (1160) |

5. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC0-inf)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: In addition, for several participants, certain PK parameter values were set to missing for the purposes of calculating descriptive statistics in the primary analysis, in accordance with the SAP. The extrapolated portion of AUC(0-inf) exceeded 20% of AUC(0-inf) in 8 participants, therefore, AUC(0-inf) was not reported for these individuals.
Measure: Mean (Standard Deviation); unit: µg.day/mL
Arm/Group | ETI-204 | Placebo
Number analyzed (Participants) | 191 | 0
µg.day/mL | 5170 (1360) |

6. Secondary Outcome: Terminal Half-life (t1/2)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: In addition, for several participants, certain PK parameter values were set to missing for the purposes of calculating descriptive statistics in the primary analysis, in accordance with the SAP. ETI-204 t1/2 values were not reported for 6 participants as they were greater than 50% of the 71-day sample collection interval.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ETI-204 | Placebo
Number analyzed (Participants) | 193 | 0
days | 20.2 (5.26) |

7. Secondary Outcome: Systemic Clearance (CL)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: In addition, for several participants, certain PK parameter values were set to missing for the purposes of calculating descriptive statistics in the primary analysis, in accordance with the SAP. The extrapolated portion of AUC(0-inf) exceeded 20% of AUC(0-inf) in 8 participants, therefore, CL was not reported for these individuals.
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | ETI-204 | Placebo
Number analyzed (Participants) | 191 | 0
Liters/day | 0.270 (0.0886) |

8. Secondary Outcome: Volume of Distribution (Vd)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: In addition, for several participants, certain PK parameter values were set to missing for the purposes of calculating descriptive statistics in the primary analysis, in accordance with the SAP. The extrapolated portion of AUC(0-inf) exceeded 20% of AUC(0-inf) in 8 participants, therefore, Vd was not reported for these individuals.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | ETI-204 | Placebo
Number analyzed (Participants) | 191 | 0
Liters | 7.41 (1.90) |

9. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: as for outcome 2
Time Frame: as for outcome 2
Population: In addition, for several participants, certain PK parameter values were set to missing for the purposes of calculating descriptive statistics in the primary analysis, in accordance with the SAP. The extrapolated portion of AUC(0-inf) exceeded 20% of AUC(0-inf) in 8 participants, therefore, Vss was not reported for these individuals.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | ETI-204 | Placebo
Number analyzed (Participants) | 191 | 0
Liters | 6.34 (1.55) |

10. Secondary Outcome: Number of Participants With Anti-ETI-204 Antibodies
Description: Serum anti-ETI-204 antibody titers were determined for all subjects in the safety population. Blood samples were collected and serum samples were assayed at an initial dilution of 1:10. Samples that were positive at the 1:10 dilution were serially diluted 1:2 and assayed until a negative result was attained. The titer of the most dilute sample yielding a positive result was recorded as the titer for that time point. Immunogenicity was measured by the number of participants in each study arm with anti-ETI-204 antibody values post-treatment ≥ 4-times higher than baseline at Day 8, 43 or 71, or if the titer was negative at baseline, the post-treatment sample(s) required a titer of at least 1:20 for it to be considered positive.
Time Frame: On Day 1 prior to the start of infusion and on Days 8, 43, and 71.
Population: All participants who received study drug and were included in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | ETI-204 | Placebo
Number analyzed (Participants) | 210 | 70
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to 71 days or 101 days (30 days after the final study visit) for subjects with ongoing adverse events at the final study visit, for each group.
Arm/Group | ETI-204 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/210 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/210 | 1/70
Other Adverse Events (participants affected / at risk) | 52/210 | 18/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETI-204 (N=210) | Placebo (N=70)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) — A 42-year old, White female was hospitalized on study Day 101 and underwent surgery for removal of both ovaries and appendix. The investigator reported an unrelated serious AE of ovarian cyst of moderate severity that resolved after one day.
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ETI-204 (N=210) | Placebo (N=70)
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 2
Infusion site erythema (General disorders) | 0 | 2
Pain (General disorders) | 3 | 2
Vessel puncture site bruise (General disorders) | 7 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 2
Urinary tract infection (Infections and infestations) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Headache (Nervous system disorders) | 21 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes